CLINICAL TRIAL: NCT03864458
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-finding Study of KHK7791 in Hyperphosphatemia Patients on Hemodialysis
Brief Title: Dose-finding Study of KHK7791 in Hyperphosphatemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7791-001
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-04

CONDITIONS: Hyperphosphatemia
Keywords: Tenapanor; Hyperphosphatemia; Hemodialysis
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- KHK7791 A (Experimental): Patients take KHK7791 low dose BID.
  Interventions: Drug: KHK7791
- KHK7791 B (Experimental): Patients take KHK7791 middle dose BID.
  Interventions: Drug: KHK7791
- KHK7791 C (Experimental): Patients take KHK7791 high dose BID.
  Interventions: Drug: KHK7791
- KHK7791 D (Experimental): Patients start at KHK7791 high dose and can down titrate weekly ,based on a GI tolerability question.
  Interventions: Drug: KHK7791
- Placebo (Placebo Comparator): Patients take Placebo BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK7791 — oral administration
  Arms: KHK7791 A; KHK7791 B; KHK7791 C; KHK7791 D
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
To evaluate the effect and safety of KHK7791 to treat Hyperphosphatemia in ptatients on HD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable chronic renal failure who have undergone hemodialysis three times per week for at least 12 weeks until screening examination.
* Dialysis conditions (dialysate, dialyzer, frequency of dialysis per week, dialysis duration, blood flow rate, and dialysate and substitution fluid flow rates), excluding dry weight, should have been unchanged during the last 2 weeks before screening examination.
* Taking phosphate binders three times per day. The prescribed drug and dosage regimen should have been unchanged during the last 4 weeks before screening examination.
* Serum phosphorus levels should be in the range of ≥3.5 and ≤6.0 mg/dL at screening examination.
* If on any vitamin D or calcimimetics regimen, then the prescribed drug and dosage regimen should have been unchanged for the last 4 weeks before screening examination.

Exclusion Criteria:

* iPTH >600 pg/mL (should be based on the most recent value from the patients' medical records, etc. before pre-enrollment)
* Having concurrent or a history of inflammatory bowel disease (IBD) or diarrhea-predominant irritable bowel syndrome
* History of gastrectomy or enterectomy (excluding endoscopic resection and cecectomy) or having undergone gastrointestinal tract surgery within 3 months before screening examination.
* Having concurrent severe heart disease [including congestive heart failure, defined as New York Heart Association (NYHA) cardiac functional classification of class III or IV, and cardiovascular disease requiring hospitalization, such as myocardial infarction] or hepatic impairment (including AST/ALT ≥100 U/L at screening examination, or cirrhosis).
* Developed cerebrovascular disease (such as cerebral infarction and hemorrhage) or cardiovascular disease (such as myocardial infarction and unstable angina) requiring hospitalization within 6 months before screening examination.
* Uncontrollable hypertension or diabetes.
* Scheduled for living donor kidney transplant, change in the mode of dialysis, home hemodialysis, or change in the dialysis center (relocate to another hospital/clinic) during the study period.
* Any diagnosis of and treatment of malignancy within 5 years before screening examination (excluding basal cell carcinoma or surgically resected intraepithelial carcinoma of uterine cervix).

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
To investigate the clinically recommended dose by comparing changes in serum phosphorus levels from baseline values at Week 6. | Week 6

SECONDARY OUTCOMES:
Changes in serum Ca × P levels from baseline. | Week 6
Changes in corrected serum calcium levels from baseline. | Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Study Site 1, Nagoya, Japan

IPD SHARING:
Plan to Share IPD: Undecided